| Statistical Analysis Plan | |
|---|---|
| Clinical Investigation Plan Title | Low-fiel <b>D</b> magn <b>E</b> ti <b>C R</b> esonance imaging of pulmonar <b>Y P</b> arenchyma changes associated wi <b>T</b> h confirmed <b>SARS-CoV-2</b> infection in children and adolescents |
| Clinical Investigation Plan Identifier | NCT04990531 |
| Clinical Investigation Plan Version | Studienprotokoll_MSOT_SMA_V2.3 on November 7 <sup>th</sup> , 2019 (Final) |
| Local Sponsor | Department of Pediatircs, University Hospital |
| | Erlangen, Friedrich-Alexander-University |
| | (FAU) Erlangen-Nürnberg |
| ocument Version SAP v1.0 (Final) | |
| Version date | 08-08-2021 |
| Confidentiality Statement | |
| All the information contained in this document is confidential. | |

# **Table of contents**

| 1. VERSION HISTORY | 3 |
|---------------------------------------------------|---|
| 2. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 3 |
| 3. Introduction | 4 |
| 4. STUDY OBJECTIVES AND ENDPOINTS | 5 |
| 5. Investigation Plan | 6 |
| 6. DETERMINATION OF SAMPLE SIZE | 7 |
| 7. TARGET PARAMETERS | 7 |
| PRIMARY TARGETS: | 7 |
| 7. STATISTICAL METHODS | 7 |
| 7.1. STUDY SUBJECTS | 7 |
| 7.2. CLINICAL INVESTIGATION PLAN (CIP) DEVIATIONS | 7 |
| 7.3 ANALYSIS SETS | 7 |
| 7.4 GENERAL METHODOLOGY | 8 |
| 7.5 HANDLING OF MISSING DATA AND DROPOUTS | 8 |
| 7.6 SAFETY EVALUATION | 8 |

# 1. Version History

| Version | Changes | Authors, Title |
|---------|--------------------|--------------------------|
| v1.0 | SAP generated | Ferdinand Knieling, M.D. |
| v.1.1 | SAP under reviewed | Biostatistician |
| | (08/08/2021) | |

# 2. List of Abbreviations and Definitions of Terms

| Abbreviation | Definition |
|--------------|------------------------------------------------------|
| SARS-CoV-2 | Severe acute respiratory syndrome coronavirus type 2 |
| COVID-19 | Survival motor neuron 2 |
| LF-MRI | Low-field magnetic resonance imaging |
| PCR | Polymerase chain reaction |

## 3. Introduction

SARS-CoV-2 (Severe acute respiratory syndrome coronavirus type 2) is a new coronavirus and identified causative agent of COVID-19 disease. They predominantly cause mild colds but can sometimes cause severe pneumonia. The long-term consequences are still largely unexplained and misunderstood, especially in children and adolescents. The aim of this study is to assess the frequency of pulmonary parenchymal changes in pediatric and adolescent patients using low-field magnetic resonance imaging (LF-MRI) in the setting of proven past SARS-CoV-2 infection.

#### 4. Study Objectives and endpoints

Determination of the frequency of lung parenchymal changes by low-field magnetic resonance imaging (LF-MRI) in past PCR-detected SARS-CoV-2 infection in pediatric and adolescent patients.

#### **Hypotheses:**

- Lung parenchymal changes in pediatric and adolescent patients with positive SARS-CoV-2 infection can be detected by LF-MRI
- The patients with changes do not show clinical symptoms

#### **Primary Objective:**

Determination of the frequency of lung parenchymal changes by LF-MRI.

#### **Secondary Goals:**

- Determination of the frequency of positive SARS-CoV-2 antibodies.
- Determination of the anamnestic frequency of clinical respiratory symptoms.

### **Endpoints**

#### **Primary Endpoint**

Frequency of lung parenchymal changes

#### **Secondary Endpoints**

Correlation of imaging results/clinical course and:

- Antibodies against SarS-CoV-2
- Physical properties of single cells: Red blood cells Deformation
- Physical properties of single cells: Red blood cells Cells size [µm³]
- Physical properties of single cells: Red blood cells Youngs modulus [kPa³]
- Physical properties of single cells: Leucocytes Deformation
- Physical properties of single cells: Leucocytes Cells size [µm³]
- Physical properties of single cells: Leucocytes Youngs modulus [kPa³]
- Physical properties of single cells: Monocytes Deformation
- Physical properties of single cells: Monocytes Cells size [µm³]
- Physical properties of single cells: Monocytes Youngs modulus [kPa³]

# 5. Investigation Plan

 This is a mono-centric, open-labeled, single arm study which aims to find the frequency of lung parenchymal changes in previous SarS-CoV-2 PCR-positive pediatric patients

- The study will include 58 patients.
- Each subject will be examined by blood samples and LF-MRI

#### **Inclusion Criteria:**

- (Past) Positive SARS-CoV-2 Infection (PCR proven)
- Age 5 to <18 years</li>

#### **Exclusion Criteria:**

- Acute SARS-CoV-2 Infection and Isolation
- Quarantine
- Pregnancy
- Critical Illness
- No consent to LF-MRI
- General contraindications for LF-MRI, such as electrical implants, pace makers, perfusion pumps)

## 6. Determination of Sample Size

With a sensitivity of 90%, specificity of 85%, precision of  $\pm 0.15$  and a prevalence of 0.3 with a confidence level of 95% for a 10% dropout, the number of cases was n=58 (including dropout).

#### 7. Target parameters

LF-MRI will be utilized to generate lung parenchymal images. Blood samples are used to assess antibody and cell properties.

**Primary Targets:** 

| Lung parencilymai changes | LF-MRT | Lung parenchymal changes |
|---------------------------|--------|--------------------------|
|---------------------------|--------|--------------------------|

## **Secondary Targets:**

| Blood sample | SARS-CoV2-Antibody |
|-------------------|-------------------------------------------|
| | Mechanical cell properties (realtime |
| | deformability cytometry) |
| | Blood count |
| Clinical Features | Age |
| (via KIS) | Gender |
| | Weight |
| | Ethnicity |
| | Time of Infection (PCR result) |
| | Interval until LF-MRT |
| | Current medication |
| | Secondary Diagnoses |
| | Symptoms during COVID (e.g cough, |
| | shortness of breath, fever) |
| | Current symptoms (e.g cough, shortness of |
| | breath, fever) |

#### 7. Statistical Methods

#### 7.1. Study Subjects

We will describe all screened and enrolled patients.

#### 7.2. Clinical Investigation Plan (CIP) Deviations

Data will be analyzed according to the SAP; any further/additional/deviation from the SAP will be reported as such. Further post-hoc analysis will be performed, if necessary.

#### 7.3 Analysis Sets

One analysis set will be created for study purpose.

#### 7.4 General Methodology

Continuous variables are given as means and standard deviations; categorical variables are provided as numbers and percentages. If appropriate, descriptive statistics will be provided using Tables.

Frequency of lung parenchymal changes will be given as percentage of total population. Clinical symptoms will be correlated to extend of changes using correlations.

As appropriate, participants will be subjected to groups (subjects with lung phenotype/subjects without lung phenotyoe): Data are tested for normal distribution using Shapiro-Wilk test prior to inferential analysis. All variables (MRI/blood values) are compared between cohorts using t-tests. If the assumption of normal distribution is violated Wilcoxon signed-rank tests is used. All inferential tests are two-tailed, p values ≤ 0.05 are considered statistically significant. Bonferroni-Holm adjustment is used to control type I error, if appropriate. All analyses are performed using GraphPad Prism (Version 7.00 or newer, GraphPad Software, La Jolla, CA, USA) and/or IBM SPSS Statistics, version 25 or newer (IBM Corp., N.Y., USA).

### 7.5 Handling of Missing Data and Dropouts

No method of imputation will be used for missing data.

#### 7.6 Safety Evaluation

During the study adverse events and serious adverse events will be monitored. The investigator is available for study subjects at any time, in case of any events.